CLINICAL TRIAL: NCT03600727
Title: Intraoperative Propofol and Dexmedetomidine on Peripheral Inflammation Induced by Hip or Knee Arthroplasty.
Brief Title: Propofol and Dexmedetomidine on Inflammation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PJ2017-06-08
Record Dates: First submitted 2018-06-27; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-04

CONDITIONS: Inflammation; Postoperative Delirium; Anesthesia
MeSH Terms: conditions — Inflammation; Emergence Delirium | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Patients receiving total hip and knee arthroplasty will be intraoperative sedated by propofol or dexmedetomidine.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor will be blinded to this study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propofol group (Experimental): Patients in this arm will be sedated by propofol.
  Interventions: Drug: Propofol
- Dexmedetomidine group (Experimental): Patients in this arm will be sedated by dexmedetomidine.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Propofol — Propofol will be used to offer intraoperative sedation for patients in Propofol group.
  Arms: Propofol group
Drug: Dexmedetomidine — Dexmedetomidine will be used to offer intraoperative sedation for patients in Dexmedetomidine group.
  Arms: Dexmedetomidine group

SUMMARY:
Dexmedetomidine, was reported to prevent postoperative delirium in elderly patients following its use in intensive care units. Possible mechanisms included improved quality of sleep and an inhibitory effect on inflammation. A greater number of studies indicated that propofol has negative effect on postoperative cognitive function. In this study, we planned to investigate the influence of these two different sedative drugs on peripheral inflammation induced by surgery and postoperative cognitive function of patients who will receive hip and knee arthroplasty.

DETAILED DESCRIPTION:
Dexmedetomidine, was reported to prevent postoperative delirium in elderly patients following its use in intensive care units. Possible mechanisms included improved quality of sleep and an inhibitory effect on inflammation. A greater number of studies indicated that propofol has negative effect on postoperative cognitive function. In this study, patients who will receive hip and knee arthroplasty will be divided to two groups: Propofol group and Dexmedetomidine group. Spinal anesthesia will be used to meet the requirement of intraoperative analgesia. Patients in two groups will be sedated by propofol and dexmedetomidine, respectively. TNF-α and IL-6 in blood will be detected. And postoperative cognitive function of patients will be investigated. The objective of this study is to clarify the influence of these two different sedative drugs on peripheral inflammation induced by surgery, and the relationship with the change of postoperative cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in this study were 65 years or older, were undergoing total hip arthroplasty, and were classified as American Society of Anesthesiologists (ASA) physical health class I-IV.

Exclusion Criteria:

* Contraindications to spinal anesthesia (i.e., coagulopathy, concurrent use of anticoagulants, infection at puncture site, and refusal of spinal anesthesia), patients with infectious diseases, patients with mental or language barriers, patients who had been anesthetized within the past 30 days, severe congestive heart failure (New York Heart Association, class IV) and/or severe chronic obstructive pulmonary disease (Global Initiative for Chronic Obstructive Lung Disease Guidelines, stages III-IV), sick sinus syndrome, severe sinus bradycardia (< 50 beats per min), and second or greater atrioventricular block without pacemaker. In addition, patients exhibiting cognitive impairment (i.e., a Mini-Mental State Examination (MMSE) score < 24) and/or preoperative delirium (i.e., positive Confusion Assessment Method (CAM) result) were excluded.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
change of the concentration of IL-6 | Preoperative and end of surgery
  Change of the concentration of plasma IL-6 from baseline to the end surgery

SECONDARY OUTCOMES:
Postoperative delirium | Postoperative (1-3 days after surgery)
  The incidence of postoperative delirium
Postoperative cognitive dysfunction | Postoperative (7 and 30 days after surgery)
  The incidence of postoperative cognitive dysfunction
change of the concentration of TNF-α | Preoperative and end of surgery
  Change of the concentration of plasma TNF-α from baseline to the end surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zhaozhao Liang, Ph.D, Study Chair — The First Affiliated Hospital of Anhui Medical University

IPD SHARING:
Plan to Share IPD: No
We don't want to open individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Memis D, Hekimoglu S, Vatan I, Yandim T, Yuksel M, Sut N. Effects of midazolam and dexmedetomidine on inflammatory responses and gastric intramucosal pH to sepsis, in critically ill patients. Br J Anaesth. 2007 Apr;98(4):550-2. doi: 10.1093/bja/aem017. No abstract available. PMID 17363413
- [Result] Shoair OA, Grasso Ii MP, Lahaye LA, Daniel R, Biddle CJ, Slattum PW. Incidence and risk factors for postoperative cognitive dysfunction in older adults undergoing major noncardiac surgery: A prospective study. J Anaesthesiol Clin Pharmacol. 2015 Jan-Mar;31(1):30-6. doi: 10.4103/0970-9185.150530. PMID 25788770